CLINICAL TRIAL: NCT02542046
Title: Uniformity of Oral Contrast Material in the Bowel
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: General Electric (Industry)
Responsible Party: Principal Investigator, Benjamin M. Yeh, MD, Professor of Radiology. Principal Investigator, University of California, San Francisco
Other Study IDs: 15-16964
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-11

CONDITIONS: Known or Suspected Abdominal Disease
MeSH Terms: interventions — Barium; Barium Sulfate; Diatrizoate; Iohexol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Barium: Patients who received barium sulfate oral contrast for abdominopelvic CT
  Interventions: Drug: Barium
- diatrizoate: Patients who received diatrizoate oral contrast for abdominopelvic CT
  Interventions: Drug: Diatrizoate
- iohexol: Patients who received iohexol oral contrast for abdominopelvic CT
  Interventions: Drug: Iohexol

INTERVENTIONS:
Drug: Barium — Administration of barium oral contrast agent prior to CT scan
  Other Names: Barium sulfate
  Groups: Barium
Drug: Diatrizoate — Administration of diatrizoate oral contrast agent prior to CT scan
  Other Names: ionic iodinated contrast agent
  Groups: diatrizoate
Drug: Iohexol — Administration of iohexol oral contrast agent prior to CT scan
  Other Names: nonionic iodinated contrast agent
  Groups: iohexol

SUMMARY:
Although positive oral contrast agents are used for the majority of abdominopelvic CT scans in the United States, the quality of bowel opacification has not been compared between the three major classes of positive oral contrast material (barium sulfate, ionic iodinated contrast material, and non-ionic iodinate contrast material). This is a retrospective single institution study of clinical records to show whether the uniformity of bowel opacification is different between the three main types of positive CT oral contrast material used in the United States (Barium sulfate, Diatrizoate, and Iohexol). The investigators will retrospectively identify 250 patients each who received oral barium sulfate, diatrizoate, and iohexol for CT scanning of the abdomen and pelvis (total 750 patients) and assess the quality of bowel lumen opacification by the positive oral contrast agents.

DETAILED DESCRIPTION:
Although positive oral contrast agents are used for the majority of abdominopelvic CT scans in the United States, the quality of bowel opacification has not been compared between the three major classes of positive oral contrast material (barium sulfate, ionic iodinated contrast material, and non-ionic iodinate contrast material). The investigators will retrospectively identify 250 patients each who received oral barium sulfate, diatrizoate, and iohexol for CT scanning of the abdomen and pelvis (total 750 patients) and assess the quality of bowel lumen opacification by the positive oral contrast agents.

Primary objective:

* To show the uniformity of bowel opacification is different between the three main types of CT oral contrast material used in the United States (Barium sulfate, Diatrizoate, and Iohexol).

Secondary objectives:

* To show whether or not one of the oral contrast agents provides more uniform opacification than the others in the proximal or distal bowel
* To assess the relative opacification of the distal small bowel (ileum) by the three contrast agents.

ELIGIBILITY:
Inclusion Criteria:

* CT scans in which oral contrast material was given

Exclusion Criteria:

* CT scans in which an obvious paucity of oral contrast material is seen,
* CT scans of patients who had studies within 1 week prior where enteric contrast may have been given, including fluoroscopic, endoscopic, or interventional studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients in our institution who had undergone CT of the Abdomen and Pelvis with administration of positive oral contrast material
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2015-09; Primary Completion 2017-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Yeh, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

REFERENCES:
- [Background] Doyle GJ, O'Donnell SC, McDonald JR, Murthy LN, Keir MJ, Wright AR. Evaluation of "Gastromiro" for bowel opacification during computed tomography: comparison with diatrizoate and barium sulphate. Br J Radiol. 1993 Aug;66(788):681-4. doi: 10.1259/0007-1285-66-788-681. PMID 7719680

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Barium | Diatrizoate | Iohexol
Started | 300 | 300 | 300
Completed | 300 | 300 | 300
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Barium | Diatrizoate | Iohexol | Total
Number analyzed (Participants) | 300 | 300 | 300 | 900
Age, Continuous [Mean (Full Range); unit: years] | 57.8 [22 to 86] | 58.9 [22 to 91] | 58.9 [21 to 90] | 58.5 [21 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 198 | 166 | 186 | 550
  Male | 102 | 134 | 114 | 350
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-uniform Bowel Lumen Opacification at CT Imaging
Description: Nonuniform contrast enhancement of the bowel lumen is a potential diagnostic pitfall at CT imaging since non-uniform enhancement may be distracting to the reader and interfere with accurate diagnosis. Conversely, homogeneously enhancing bowel lumen makes it easier to assess the bowel for potential disease. For each patient's CT scan, the bowel that is seen to be visibly opacified by oral contrast at CT imaging will be assessed as a whole as showing the presence or absence of nonuniform contrast enhancement of the lumen.
Time Frame: within 1 day from administration of oral contrast. The CT scan generally occurs within 3 hours after oral contrast administration, and the CT scan images will be evaluated for the imaging appearance of oral contrast uniformity for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Barium | Diatrizoate | Iohexol
Number analyzed (Participants) | 300 | 300 | 300
Participants | 140 | 73 | 68

2. Primary Outcome: Severity of CT Imaging Artifacts Caused by the Oral Contrast Agent
Description: For the segments of bowel visibly opacified by oral contrast, the severity of CT imaging artifacts caused by the oral contrast agent was recorded on the following 3 point scale: 0 = no artifact; 1 = mild artifact without impairment of anatomic delineation; 2 = severe artifact with impairment of anatomic delineation. Lower scores are preferred
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Barium | Diatrizoate | Iohexol
Number analyzed (Participants) | 300 | 300 | 300
Participants
  No artifact | 296 | 294 | 296
  Mild artifact | 4 | 6 | 4
  Severe artifact | 0 | 0 | 0

3. Secondary Outcome: Extent of Bowel Opacification of Bowel at CT Imaging
Description: The most distal segment of bowel (stomach, jejunum, ileum, and /or colon) that was opacified by contrast material at the time of CT imaging was recorded
Time Frame: within 1 day from administration of oral contrast. The CT scan generally occurs within 3 hours after oral contrast administration, and the CT scan images will be evaluated for imaging appearance of oral contrast seen in bowel for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Barium | Diatrizoate | Iohexol
Number analyzed (Participants) | 300 | 300 | 300
Participants
  Stomach | 0 | 0 | 0
  Duodenum | 2 | 0 | 0
  Jejunum | 24 | 27 | 40
  Ileum | 169 | 174 | 226
  Colon | 105 | 99 | 34

ADVERSE EVENTS:
Arm/Group | Barium | Diatrizoate | Iohexol
All-Cause Mortality (participants affected / at risk) | 0/300 | 0/300 | 0/300
Serious Adverse Events (participants affected / at risk) | 0/300 | 0/300 | 0/300
Other Adverse Events (participants affected / at risk) | 0/300 | 0/300 | 0/300

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No